CLINICAL TRIAL: NCT01760304
Title: Evaluation of Changes in Cardiac Function in COPD Patients With Resting Hyperinflation After Administration of Budesonide/Formoterol (Symbicort®) Compared With Placebo
Brief Title: Changes in Cardiac Function in COPD Patients After Administration of Budesonide/Formoterol (Symbicort®) Versus Placebo
Acronym: AZCO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decided to stop the study due to expiration of blinded placebo .
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Bartolome Celli, Lecturer in Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-P-001576/1; D589BL00021/ISSSYMB0033 (Other Grant/Funding Number: AstraZeneca pharmaceuticals)
Record Dates: First submitted 2012-10-23; First posted 2013-01-04 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide / Formoterol (Experimental): This is a crossover study, where every patient will receive in a blinded fashion either Budesonide/Formoterol (Symbicort ® ) or placebo
  Interventions: Drug: Budesonide / Formoterol
- Placebo (Placebo Comparator): This is a crossover study, where every patient will receive in a blinded fashion either Budesonide/Formoterol (Symbicort ® ) or placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide / Formoterol — Budesonide/ formoterol (B/F) 160/4.5 mcg per activation. Subject who met inclusion criteria will be have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of either Budesonide/formoterol (B/F) 160/4.5 mcg per activation (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
  Other Names: Symbicort ®
  Arms: Budesonide / Formoterol
Drug: Placebo — Each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of placebo (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
  Arms: Placebo

SUMMARY:
To investigate whether Budesonide/Formoterol (Symbicort ®) therapy can improve heart function at rest by decreasing lung hyperinflation in patients with COPD (Chronic Obstructive Pulmonary Disease).

DETAILED DESCRIPTION:
Patients with moderate to advanced COPD are known to have static hyperinflation (at rest) as a consequence of expiratory flow limitation. Hyperinflation is easily detected by measuring lung volumes during standard pulmonary function testing.

Decreased Inspiratory Capacity (IC) secondary to hyperinflation has been described as a predictor of mortality in COPD, and as a limiting factor for the maximal tidal volume attained during exercise. Hyperinflation has been linked to a low cardiac output in part by limiting left ventricular ejection fraction during exercise.

Treatment with inhaled anticholinergic agents or long-acting beta agonists (LABA) and combination of the LABA formoterol and budesonide has been shown to improve IC and decrease lung hyperinflation. Bronchodilators have been shown to improve exercise endurance in COPD when combined with pulmonary rehabilitation, however the exact mechanism: improvement of lung mechanics and /or improvement in cardiac function is not well known.

Impedance cardiography (ICG) has emerged as a method to measure cardiac output without the need for invasive devices. Cardiac output measurement by impedance cardiography (CO-ICG) is a valid and reproducible method. It has been shown to have good correlation with thermodilution and the direct Fick method for the measurement of stroke volume and cardiac output.

In addition, the oxygen pulse, easily obtained by dividing the measured oxygen uptake by the heart rate (VO2/HR) provides an adequate reflection of cardiac stroke volume when the systemic extraction of oxygen is stable.

This method has been used to evaluate the effect of static and dynamic hyperinflation on cardiac function.

This pilot study is designed to be a single center (Brigham and Women's Hospital), randomized, placebo-controlled, double blind, crossover study of 14 patients (male and female 40 to 80 years old) with COPD and static hyperinflation.

The primary endpoint is the measurement of stroke volume, cardiac output and oxygen pulse at rest before and after the administration of budesonide/formoterol compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Outpatients subjects of either sex between ages 40-80 years, with a diagnosis of COPD. COPD will be characterized as the presence of airflow obstruction with an FEV1/FVC < 0.7 (Forced Expiratory Volume at one second / Forced Vital Capacity) and a FEV1 (Forced Expiratory Volume at one second ) 80% of predicted. All patients must have lung hyperinflation as demonstrated by an increase of ≥100 ml after the administration of budesonide/formoterol. All patients must have a cigarette smoking history of more than 10 pack-years, and be able to perform all the specified procedures as required by the protocol.

Exclusion Criteria:

1. Patients with other significant diseases (recent < 6 weeks COPD exacerbation) that could place the patient at risk because of participation in the study, or which may influence the results of the study or the patients' ability to participate in the study.
2. All patients with a recent (<1 year) history of myocardial infarction, or with a recent history of heart failure (NYHA class III and IV, pulmonary edema, or patients with cardiac arrhythmias.
3. Patients on daytime oxygen therapy.
4. Patients with known active tuberculosis.
5. Patients with a history of active cancer except for non-metastatic skin cancer.
6. Patients who have undergone thoracotomy, sternotomy, major cardiopulmonary intervention (lung resection, open heart surgery, etc), or other procedure in the 6 months prior to evaluation likely to cause instability of pulmonary status.
7. Patients with upper respiratory infection in the past six weeks.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bartolome R Celli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide / Formoterol , Then Placebo: This is a crossover study, where every patient signed to this arm received in a blinded fashion Budesonide/Formoterol (Symbicort ® ) 160/4.5 mcg (2 inhalations) then placebo
  Budesonide / Formoterol: Budesonide/ formoterol (B/F) 160/4.5 mcg per activation.
  Subject who met inclusion criteria will be have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of Budesonide/formoterol (B/F) 160/4.5 mcg per activation (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
- Placebo Then Budesonide/Formoterol: Every patient in this arm received in a blinded fashion placebo first then Budesonide/Formoterol (Symbicort ® )
  Placebo: Each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of placebo (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
Period: Overall Study
Arm/Group | Budesonide / Formoterol , Then Placebo | Placebo Then Budesonide/Formoterol
Started (This is a double crossover study design, therefore each patient use intervention and placebo) | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Budesonide / Formoterol First , Then Placebo: Subjects received in a blinded fashion Budesonide/Formoterol (Symbicort ® )2 inhalations (160/4.5) then placebo 2 inhalations Budesonide / Formoterol: Budesonide/ formoterol (B/F) 160/4.5 mcg per activation.
  Subject will have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs Budesonide/formoterol (B/F) 160/4.5 mcg per activation (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
- Placebo First, Then Budesonide/Formoterol: Subjects received in a blinded fashion placebo 2 inhalation then Budesonide/Formoterol (Symbicort ® )2 inhalations (160/4.5)
  Subject will have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs Placebo on visit 1 then Budesonide/formoterol (B/F) 160/4.5 msg per activation on visit 2 (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
- Total: Total of all reporting groups
Arm/Group | Budesonide / Formoterol First , Then Placebo | Placebo First, Then Budesonide/Formoterol | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7) | 70 (10) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output
Description: Impedance cardiography (ICG) (BioZ Dx ICG machine, by CardioDynamics) was used to measure cardiac output without the need for invasive devices. Cardiac output measurement by impedance cardiography (CO-ICG) is a plethysmography technique using sensors to detect the properties of the blood flow in the thorax.
  All subjects had on each visit a baseline measurement at rest and then 45 minutes after intervention (Budesonide/formoterol or Placebo). Measurement were performed at rest for 5 minutes to obtain a steady state and the last 2 minutes were taken for analysis as an averaged value labeled as pre and post intervention. For the analysis we calculated the difference from pre and post intervention at each visit. Paired t-test was used to compare the mean+/- SD of the pre and post difference when taking the study drug vs placebo.
Time Frame: Change from Baseline and at 45 minutes after administration of study medication or placebo
Measure: Mean (95% Confidence Interval); unit: ml/beat
Groups:
- Budesonide / Formoterol: In this arm patients received in a blinded fashion Budesonide/Formoterol (Symbicort ® ) first then placebo on subsequent visit (cross-over study)
  Budesonide / Formoterol: Budesonide/ formoterol (B/F) 160/4.5 mcg per activation.
  Subject who met inclusion criteria will have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of Budesonide/formoterol (B/F) 160/4.5 mcg per activation (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
- Placebo: In this arm patients received in a blinded fashion placebo first then Budesonide/Formoterol (Symbicort ® ) on subsequent visit (cross-over study).
  Placebo: On visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of placebo (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
Arm/Group | Budesonide / Formoterol | Placebo
Number analyzed (Participants) | 5 | 5
ml/beat | -0.1 [-1.1 to 0.8] | 1.9 [1.3 to 2.5]
Statistical Analysis 1: Comparison: Budesonide / Formoterol; a paired t-test was calculated comparing baseline measures and post intervention; Test type: Superiority; p = 0.769, 2-sided paired t-test
Statistical Analysis 2: Comparison: Placebo; a paired t-test was calculated comparing baseline measures and post intervention; Test type: Superiority or Other; p < 0.0001, paired T-test

2. Secondary Outcome: Lung Hyperinflation
Description: Evaluation of lung hyperinflation as determined by Pulmonary function test where Inspiratory Capacity (IC) before and 45 minutes after the administration of the budesonide/formoterol or placebo.
Time Frame: Change from Baseline and after 45 minutes after administration of study medication or placebo
Measure: Mean (95% Confidence Interval); unit: Liters
Groups:
- Budesonide / Formoterol: In this arm patients received in a blinded fashion Budesonide/Formoterol (Symbicort ® ) first then placebo on subsequent visit (cross-over study)
  Budesonide / Formoterol: Budesonide/ formoterol (B/F) 160/4.5 mcg per activation.
  Subject who met inclusion criteria will be have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of either Budesonide/formoterol (B/F) 160/4.5 mcg per activation (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
- Placebo: In this arm patients will received in a blinded fashion placebo first then Budesonide/Formoterol (Symbicort ® ) on subsequent visit (cross-over study)
  Placebo: Each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of placebo (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
Arm/Group | Budesonide / Formoterol | Placebo
Number analyzed (Participants) | 5 | 5
Liters | 0.34 [0.166 to 0.514] | -0.058 [-0.234 to 0.118]

3. Secondary Outcome: Evaluation of O2 Pulse
Description: Evaluation of O2 Pulse is the measurement of oxygen consumption pre and post intervention
Time Frame: Change from Baseline and 45 minutes after administration of study medication or placebo
Measure: Mean (95% Confidence Interval); unit: ml/beat
Groups:
- Budesonide / Formoterol: This is a crossover study, where every patient will receive in a blinded fashion either Budesonide/Formoterol (Symbicort ® ) or placebo
  Budesonide / Formoterol: Budesonide/ formoterol (B/F) 160/4.5 mcg per activation.
  Subject who met inclusion criteria will be have at each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of either Budesonide/formoterol (B/F) 160/4.5 mcg per activation (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
- Placebo: This is a crossover study, where every patient will receive in a blinded fashion either Budesonide/Formoterol (Symbicort ® ) or placebo
  Placebo: Each visit day lung function, heart function and breathlessness measurements at baseline, then they will receive 2 puffs of placebo (as per the randomization-crossover schema).
  After 45 minutes , the above measurements will be repeated.
Arm/Group | Budesonide / Formoterol | Placebo
Number analyzed (Participants) | 5 | 5
ml/beat | -0.03 [-0.10 to 0.03] | 0.17 [0.08 to 0.26]
Statistical Analysis 1: Comparison: Budesonide / Formoterol vs Placebo; Test type: Superiority or Other; p < 0.05, paired t-test

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Budesonide / Formoterol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No